CLINICAL TRIAL: NCT01924819
Title: A Randomised Phase II/III Trial of Preoperative Chemoradiotherapy Versus Preoperative Chemotherapy for Resectable Gastric Cancer
Brief Title: Trial of Preoperative Therapy for Gastric and Esophagogastric Junction Adenocarcinoma
Acronym: TOPGEAR
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Australasian Gastro-Intestinal Trials Group (Network)
Collaborators: National Health and Medical Research Council, Australia (Other); Trans Tasman Radiation Oncology Group (Other); European Organisation for Research and Treatment of Cancer - EORTC (Network); NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG0407GR; ACTRN12609000035224 (Registry Identifier: ANZCTR); U1111-1146-0762 (Other: Universal Trial Number); TROG 08.08 (Other: TROG); 22114-40111 (Other: EORTC); GA.1 (Other: NCIC CTG)
Record Dates: First submitted 2013-08-14; First posted 2013-08-19 (Estimated); Last update posted 2025-03-04 (Actual); Status verified 2024-08

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; Stomach cancer; Chemoradiotherapy; Surgery; Chemotherapy; Neoadjuvant
MeSH Terms: conditions — Stomach Neoplasms | interventions — Epirubicin; Cisplatin; Fluorouracil; Capecitabine; Oxaliplatin; Leucovorin; Docetaxel; Gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preoperative chemoradiotherapy (Experimental): 2 cycles preoperative chemotherapy with: epirubicin + cisplatin + 5-fluorouracil. (5-fluorouracil may be replaced with capecitabine).
  OR epirubicin + oxaliplatin + capecitabine OR 3 cycles of 5-fluorouracil +Leucovorin + oxaliplatin + docetaxel
  5 weeks preoperative chemoradiotherapy.
  Gastric resection.
  3 cycles adjuvant chemotherapy with: epirubicin + cisplatin + 5-fluorouracil. (5-fluorouracil may be replaced with capecitabine).
  OR epirubicin + oxaliplatin + capecitabine OR 4 cycles of 5-fluorouracil +Leucovorin + oxaliplatin + docetaxel
  Interventions: Drug: Epirubicin + cisplatin + 5-fluorouracil OR epirubicin + cisplatin + capecitabine OR epirubicin + oxaliplatin + capecitabine OR 5-Fluorouracil + leucovorin + oxaliplatin + docetaxel; Radiation: Preoperative chemoradiotherapy; Procedure: Gastric resection
- Preoperative chemotherapy (Active Comparator): 3 cycles preoperative chemotherapy with: epirubicin + cisplatin + 5-fluorouracil. (5-fluorouracil may be replaced with capecitabine).
  OR epirubicin + oxaliplatin + capecitabine OR 4 cycles of 5-fluorouracil +Leucovorin + oxaliplatin + docetaxel
  Gastric resection.
  3 cycles adjuvant chemotherapy with: epirubicin + cisplatin + 5-fluorouracil. (5-fluorouracil may be replaced with capecitabine) OR epirubicin + oxaliplatin + capecitabine OR 4 cycles of 5-fluorouracil +Leucovorin + oxaliplatin + docetaxel
  Interventions: Drug: Epirubicin + cisplatin + 5-fluorouracil OR epirubicin + cisplatin + capecitabine OR epirubicin + oxaliplatin + capecitabine OR 5-Fluorouracil + leucovorin + oxaliplatin + docetaxel; Procedure: Gastric resection

INTERVENTIONS:
Drug: Epirubicin + cisplatin + 5-fluorouracil OR epirubicin + cisplatin + capecitabine OR epirubicin + oxaliplatin + capecitabine OR 5-Fluorouracil + leucovorin + oxaliplatin + docetaxel — Epirubicin 50 mg/m2 IV day 1, cisplatin 60 mg/m2 IV day 1, 5-fluorouracil 200 mg/m2/d IV 21 day continuous infusion (ECF chemotherapy).
  Epirubicin 50 mg/m2 IV day 1, Cisplatin 60 mg/m2 IV day 1, Capecitabine (X = Xeloda) 625mg/m2, bid days 1-21 (ECX chemotherapy)
  Epirubicin 50mg/m2 IV day 1, Oxaliplatin (O) 130mg/m2 IV day 1, Capecitabine 625mg/m2, bid days 1-21 (EOX chemotherapy)
  5-Fluorouracil 2600 mg/m² IV 24 h infusion day 1, Leucovorin (L) 200 mg/m² IV day 1, Oxaliplatin 85 mg/m² IV day 1, Docetaxel (T) 50 mg/m² IV day 1 (FLOT chemotherapy)
  Other Names: Epirubicin hydrochloride, Pharmorubicin, Ellence; Platinol; 5-FU, Adrucil, Carac, Efudex. Efudix; Xeloda; Eloxatin; Folinic acid, 5-formyl tetrahydrofolic acid, Citrovorum Factor; Taxotere, Docetere
Radiation: Preoperative chemoradiotherapy — Chemotherapy: Continuous infusional 5-fluorouracil 200mg/m2/day, 7 days per week, throughout the entire period of radiotherapy or capecitabine 825 mg/m2, oral tablet twice daily, days 1-5 of each week of radiotherapy (without weekends).
  Radiotherapy: 45 Gy of radiation in 25 fractions, five days per week for five weeks.
  Arms: Preoperative chemoradiotherapy
Procedure: Gastric resection — The acceptable resections are a total gastrectomy, a subtotal gastrectomy, and an esophagogastrectomy (Ivor-Lewis esophagogastrectomy for gastroesophageal junction cancers [Siewert Type II and Siewert Type III] invading up to but no more than 2cm of the lower esophagus). The minimum extent of the operation should be a D1+ lymph node dissection but it is recommended that a D2 dissection be performed or a D1+ for gastroesophageal junction cancers requiring an esophagogastrectomy.

SUMMARY:
Gastric cancer remains a significant global public health problem. Although in developed countries its incidence has dramatically decreased, on a worldwide scale it is still a leading cause of cancer-related deaths. Surgery is the only potentially curative treatment for gastric cancer. Although the survival rates for patients with early stage disease (stage 1A and 1B) are good, this subgroup of patients constitutes only 20% of those undergoing resection. The majority of patients will have locally advanced or metastatic disease at presentation, which has an extremely poor prognosis. The current five-year survival rate for gastric cancer in Western countries is approximately 20-30%, a figure that has improved little over the past 30 years. The intervention arm in TOPGEAR consists of pre-operative chemotherapy, pre-operative chemoradiotherapy, surgery and post-operative chemotherapy. The control arm consists of pre-operative chemotherapy, surgery and post-operative chemotherapy. The primary objective of TOPGEAR is to investigate whether the addition of chemoradiotherapy to chemotherapy is superior to chemotherapy alone in the neoadjuvant setting by improving pathological complete response rates in the first instance, and subsequently overall survival, in patients undergoing adequate surgery (D1+ dissection) for resectable gastric cancer.

DETAILED DESCRIPTION:
Purpose:

The purpose of this phase II/III clinical trial is to determine if pre-operative chemoradiotherapy improves overall survival in participants with resectable gastric cancer.

Trial details:

Participants will be randomised to receive either pre-operative chemotherapy or pre-operative chemoradiotherapy. The will undergo surgery and then receive further post-operative chemotherapy. Participants will be followed up for 5 years after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the stomach or gastroesophageal junction (GEJ) that is:

  1. Stage IB (T1N1 only, T2N0 not eligible) - IIIC, i.e. T3 - T4 and/or node positive, according to American Joint Committee on Cancer (AJCC) 7th edition.
  2. Considered operable following initial staging investigations (surgeon believes that an R0 resection can be achieved) (GEJ tumours are defined as tumours that arise in the cardia or at the GEJ that do not involve more than 2cm of the lower esophagus, i.e. Siewert Type II and Siewert Type III)
* Age >=18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Adequate organ function defined as follows:

  1. Bone marrow: Haemoglobin >=90 g/L, Absolute neutrophil count (ANC) >=1.5 x 10⁹ /L, White blood cell count >=3 x 10⁹ /L, Platelet count >=100 x 10⁹ /L
  2. Hepatic: Serum bilirubin <=1.5 x upper limit of normal (ULN), aspartate aminotransferase (AST) and/or alanine transaminase (ALT) <=3.0 x ULN
  3. Renal: Serum creatinine <=0.150 mmol/L, Calculated creatinine clearance >=50 mL/min
* Disease which can be radically treated with radiotherapy to 45 Gy with standard fractionation
* Any patient with a history of ischaemic heart disease and abnormal ECG, or who is over 60 years of age should have a pre-treatment evaluation of cardiac function with a multigated acquisition (MUGA) scan or echocardiogram. Patients will only be included if the left ventricular ejection fraction is >=50%.
* Written informed consent obtained before randomization
* Negative pregnancy test for women of childbearing potential within 7 days of commencing study treatment. Males and females of reproductive potential must agree to practice adequate contraceptive measures.

Exclusion Criteria:

* Evidence of metastatic disease
* Prior chemotherapy or radiotherapy
* Patients with a past history of cancer in the 5 years before randomization except for the following. Patients with squamous or basal cell carcinoma of the skin that has been effectively treated, and patients with carcinoma in situ of the cervix that has been treated by operation only are eligible, even if they were diagnosed and treated within the 5 years before randomization.
* Patients with other significant underlying medical conditions that may be aggravated by the study treatment or are not controlled
* Pregnant or lactating females or female patients of childbearing potential who have not been surgically sterilized or are without adequate contraceptive measures
* Cardiac failure and other contraindications to epirubicin
* Patients with impaired gastrointestinal absorption for whatever reason
* Patients medically unfit for cisplatin chemotherapy due to one or more of the following reasons:

  1. Clinically significant sensorineural hearing impairment (audiometric abnormalities without corresponding clinical deafness will not be regarded as a contraindication to cisplatin)
  2. Severe tinnitus
  3. Renal impairment (GFR <=50ml/min)
  4. Peripheral neuropathy >=grade 2
  5. Inability to tolerate intravenous hydration e.g due to cardiac disease
  6. Co-morbidities (based on clinical judgement by the investigator) that in the view of the investigator would preclude the safe administration of cisplatin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 574 (Actual)
Dates: Start 2009-09; Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Up to 5 years
  The interval from the date of randomisation to the date of death from any cause, or the date last known alive.

SECONDARY OUTCOMES:
Disease free survival | Up to 5 years
  The time from the date of randomisation to the first observation of disease progression or death due to any cause.
Pathological response rate | At time of surgery
  The extent of reduction in tumour size following pre-operative treatment, as determined by macroscopic and microscopic assessment of the tumour.
Proportion of participants with given grades of toxicities | Up to 5 years
  The proportion of participants starting at least one cycle of treatment and the grades of the toxicities reported.
Surgical complete resection rate (R0) | At the time of surgery
  The complete macroscopic resection of gross tumour with negative surgical margins.

CONTACTS AND LOCATIONS:
Overall Officials: Trevor Leong, MBBS, MD, Study Chair — Peter MacCallum Cancer Centre, Australia
Locations (59):
- Australia (21):
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Chris O Brien Lifehouse, Sydney, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - Nepean Hospital, Sydney, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - St George Hospital, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - The Tweed Hospital, Tweed Heads, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Flinders Medical Centre, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Launceston General Hospital, Launceston, Tasmania
  - Geelong Hospital, Geelong, Victoria
  - Austin Hospital, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - St Vincent's Hospital, Melbourne, Victoria
  - Sunshine Hospital (Western Health), Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Belgium (7):
  - AZ Klina, Brasschaat
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Hospital De Jolimont, La Louvière
  - U.Z Leuven Campus Gasthuisberg, Leuven
  - AZ Damiaan, Ostend
  - AZ Turnhout- Campus Sint Elisabeth, Turnhout
  - Centre Hospitalier Peltzer- La Tourelle, Verviers
- Canada (15):
  - BCCA - Vancouver Centre, Vancouver, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Grand River Regional Cancer Center, Kitchener, Kitchener, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Health Research Institute, Ottawa, Ontario
  - Odette Cancer Centre, Sunnybrook Hospital, Toronto, Ontario
  - UHN - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Hospital Notre-Dame, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Charles University Hospital, Hradec Králové, Czechia
- France (4):
  - Institut Sainte Catherine, Avignon
  - CHRU de Besancon Hopital Jean Minjoz, Besançon
  - Centre Hospitalier de Belfort Montbeliard site du Mittan, Montbéliard
  - Centre Paul Strauss, Strasbourg
- Klinikum der Universitaet Muenchen - Campus Grosshadern, München, Bavaria, Germany
- Israel (2):
  - Rambam Medical Center, Haifa
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- New Zealand (3):
  - Auckland Hospital, Auckland
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton
- The Institute of Oncology, Ljubljana, Slovenia
- Spain (4):
  - ICO L Hospitalet Hospital Duran i Reynals (Institut Catala D Oncologia), L'Hospitalet de Llobregat, Barcelona
  - Institut Catala d Oncologia - ICO Badalona - Hospital Germans Trias i Pujol, Badalona
  - Vall D Hebron University Hospital, Barcelona
  - Hospital Clinico Universitario De Valencia, Valencia

REFERENCES:
- [Derived] Leong T, Smithers BM, Michael M, Haustermans K, Wong R, Gebski V, O'Connell RL, Zalcberg J, Boussioutas A, Findlay M, Willis D, Moore A, Murray WK, Lordick F, O'Callaghan C, Swallow C, Darling G, Miller D, Strickland A, Liberman M, Mineur L, Simes J; Australasian Gastro-Intestinal Trials Group, National Health and Medical Research Council Clinical Trials Centre, Trans-Tasman Radiation Oncology Group, European Organisation for Research and Treatment of Cancer, and Canadian Cancer Trials Group. Preoperative Chemoradiotherapy for Resectable Gastric Cancer. N Engl J Med. 2024 Nov 14;391(19):1810-1821. doi: 10.1056/NEJMoa2405195. Epub 2024 Sep 14. PMID 39282905